CLINICAL TRIAL: NCT05685238
Title: Open-label, Long-term Safety and Efficacy Study of Mim8 in Participants With Haemophilia A With or Without Inhibitors
Brief Title: A Research Study Looking at Long-term Treatment With Mim8 in People With Haemophilia A (FRONTIER 4)
Acronym: FRONTIER4
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN7769-4532; U1111-1274-4426 (Other: World Health Organization (WHO)); 2022-502215-10 (EudraCT Number)
Record Dates: First submitted 2023-01-04; First posted 2023-01-17 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Haemophilia A; Haemophilia A With Inhibitors
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Experimental): Participants entering from the multiple ascending dose (MAD) part of study NN7769-4513. In part 1, participants will receive Mim8 prophylaxis (PPX) subcutaneous (s.c.) administration using enhanced cartridge for 26 weeks. In part 2, participants will receive Mim8 PPX s.c. administration using enhanced cartridge or DV3407 pen-injector once it is approved.
  Interventions: Drug: Mim8
- Arm 2 (Experimental): Participants entering from study NN7769-4514, NN7769-4728 and NN7769-4516. In part 1, participants will receive Mim8 PPX s.c. administration using DV3407 pen-injector for 26 weeks. In part 2, participants will receive Mim8 PPX s.c. administration using DV3407 pen-injector.
  Interventions: Drug: Mim8
- Arm 3 (Experimental): In part 1 and 2, participants will receive Mim8 PPX s.c. administration using DV3407 pen-injector.
  Interventions: Drug: Mim8

INTERVENTIONS:
Drug: Mim8 — Participants in arm 1 will administer Mim8 using an enhanced cartridge and switch to the DV3407 pen-injector once it is approved. Participants in arm 2 and 3 will use the DV3407 pen injector.

SUMMARY:
This study is looking at how Mim8 works in people with haemophilia A, who either have inhibitors or do not have inhibitors. Mim8 is a new medicine that will be used to avoid bleeding episodes. Mim8 works by replacing the function of the missing clotting factor VIII (FVIII). The study will last for up to 5.5 years. The duration of the study depends on when the participant enrolled in this study. The study will end if Mim8 is approved and marketed in participant's country during the study, or the study will end in June 2028, whichever comes first. Participants will get up to 262 injections; the number of injections depends on how often participants will get injections and how long time participants take part in the study. While taking part in this study, there are some restrictions about what medicine participants can use. The study doctor will tell the participants more about this. In case the participants experience bleeds, these can be treated with additional haemostatic medicine as agreed with the study doctor. Female participants cannot take part if they are pregnant, breast-feeding or plan to get pregnant during the study period.

ELIGIBILITY:
Arm 1 & 2:

Inclusion Criteria:

1. Informed consent obtained before any study related activities. Study related activities are any procedures that are carried out as part of the study, including activities to determine suitability for the study.
2. Male or female with diagnosis of congenital haemophilia A based on medical records.
3. Ongoing participation in study NN7769-4513, NN7769-4514, NN7769-4516, or NN7769-4728 at the time of transfer. Participant should qualify either of the following criteria:

   1. Participant from study NN7769-4513, who has participated in the extension part of the study for at least 12 weeks prior to enrolment in study NN7769-4532, or,
   2. Participant has completed the end of treatment visit for study NN7769-4514, NN7769-4516 or NN7769-4728.
4. Participant and/or participant's parent(s)/participant's Legally acceptable representative (LAR) willingness and ability to comply with scheduled visits and study procedures, including the completion of diary.

Exclusion Criteria:

1. Any disorder, except for conditions associated with haemophilia A, which in the investigator's opinion might jeopardise participant's safety or compliance with the protocol.
2. Participant who has discontinued or been withdrawn from studies NN7769-4513, NN7769-4514, NN7769-4516, or NN7769-4728.
3. Previous participation in this study. Participation is defined as signed informed consent.
4. Female who is pregnant, breast-feeding or intends to become pregnant.
5. Female of child-bearing potential and not using a highly effective contraceptive method (highly effective contraceptive measures or as required by local regulation or practice).
6. Participation (i.e., signed informed consent) in any interventional, clinical study (except from study NN7769-4513, NN7769-4514, NN7769-4516, or NN7769-4728) of an approved or non-approved investigational medicinal product.
7. Any planned major surgery, during part 1 of the study.
8. Mental incapacity, unwillingness to cooperate, or a language barrier precluding adequate understanding and cooperation.

Arm 3:

Inclusion criteria

1. Informed consent obtained before any study-related activities. Study-related activities are any procedures that are carried out as part of the study, including activities to determine suitability for the study.
2. Male or female with diagnosis of congenital severe haemophilia A (endogenous FVIII activity less than (<) 1 percentage [%]) with or without FVIII inhibitors based on medical records.
3. Aged <1 year at the time of signing informed consent.
4. Body weight greater than or equal to (≥) 3.2 kilograms at the time of signing informed consent.
5. previously untreated patients (PUPs) or minimally treated patients (MTPs) (i.e., up to 5 days of exposure to haemophilia-related treatment such as plasma-derived FVIII, recombinant FVIII, fresh frozen plasma, cryoprecipitate, or whole blood products).
6. Full-term pregnancy (gestational age ≥37 weeks).
7. Participant's parent(s)/LAR(s) willingness and ability to comply with scheduled visits and Arm 3 (infant) procedures, including the completion of diary and patient reported outcome (PRO) questionnaire.
8. Participants <3 months of age must show no signs of active intracranial haemorrhage at screening. This is confirmed by cranial ultrasound performed according to local practice and regardless of delivery method.
9. Receipt of vitamin K prophylaxis (as per local standard practice).
10. Availability of historical results in medical records for:

    a. activated partial thromboplastin time (aPTT) b. FVIII levels.
11. Availability of historical results in medical records or pre-dose sample taken for:

    1. fibrinogen
    2. haematology parameters
    3. biochemistry parameters (aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT), bilirubin and creatinine).

Exclusion criteria

1. Known or suspected hypersensitivity to trial product or related products.
2. Previous participation in study 4532. Participation is defined as signed informed consent.
3. Participation (i.e., signed informed consent) in any interventional clinical study with receipt of the last dose within 6 months (or 5 half-lives of the investigational medicinal product, whichever is shorter) before planned enrolment.
4. Exposure to non-factor haemostatic products for bleeding prophylaxis within 6 months (or 5 half-lives of the medicinal product, whichever is shorter) before planned enrolment.
5. Known congenital or acquired coagulation disorders other than haemophilia A.
6. Other conditions (e.g., autoimmune disease) or laboratory abnormality that may increase the risk of bleeding or thrombosis, as evaluated by the investigator. Any disorder, except for conditions associated with haemophilia A, that in the investigator's opinion might jeopardise the participant's safety or compliance with the protocol.

8. Lack of adequate parental/legally acceptable representative (LAR) support to enter accurately and timely information regarding treatment and bleeding episodes into an (electronic) diary.

9. Previous or current treatment for thromboembolic disease (with the exception of previous catheter-associated thrombosis for which anti-thrombotic treatment is not currently ongoing) or signs of thromboembolic disease.

10. Any planned major surgery, during part 1 of Arm 3 (infant). For definition of major surgery.

11. Immune tolerance induction planned to take place after treatment initiation.

12. Hepatic dysfunction defined as AST and/or ALT greater than (>) 3 times the upper limit of normal (ULN) combined with total bilirubin >1.5 times the ULN.

13. Serum creatinine above 1.5 times the ULN.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 451 (Estimated)
Dates: Start 2023-02-13 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Arm 1 and 2: Number of treatment emergent adverse events | From week 0 until end of study (up to 283 weeks)
  Measured as count of events.
Arm 3: Number of treatment emergent adverse events | From treatment initiation (week 0) until end of study (up to 124 weeks)
  Measured as count of events.

SECONDARY OUTCOMES:
Arm 1 and 2: Number of injection site reactions | From week 0 until end of treatment (up to 262 weeks)
  Measured as count of reactions.
Arm 1 and 2: Occurrence of anti Mim8 antibodies | From week 0 until end of treatment (up to 262 weeks)
  Measured as count of participants.
Arm 1 and 2: Number of treated bleeding episodes | From week 0 until end of treatment (up to 262 weeks)
  Measured as count of bleeds.
Arm 1 and 2: Number of treated spontaneous bleeding episodes | From week 0 until end of treatment (up to 262 weeks)
  Measured as count of bleeds.
Arm 1 and 2: Number of treated traumatic bleeding episodes | From week 0 until end of treatment (up to 262 weeks)
  Measured as count of bleeds.
Arm 1 and 2: Number of treated joint bleeding episodes | From week 0 until end of treatment (up to 262 weeks)
  Measured as count of bleeds.
Arm 2: Number of treated target joint bleeding episodes | From week 0 until end of treatment (up to 262 weeks)
  Measured as count of bleeds.
Arm 1 and 2: Mim8 plasma concentration | From week 0 until end of treatment (up to 262 weeks)
  Measured as micrograms per milliliter (µg/mL).
Arm 2: Device handling using haemophilia device assessment tool (HDAT) (applicable for participants in arm 2 only) | From week 26 until end of treatment (up to 262 weeks)
  Measured as percentage of participants.
Arm 3: Number of injection site reactions | From treatment initiation (week 0) until end of treatment (up to 103 weeks)
  Measured as count of reactions.
Arm 3: Occurrence of anti Mim8 antibodies | From treatment initiation (week 0) until end of treatment (up to 103 weeks)
  Measured as count of participants.
Arm 3: Number of treated bleeding episodes | From treatment initiation (week 0) until end of treatment (up to 103 weeks)
  Measured as count of bleeds.
Arm 3: Number of treated spontaneous bleeding episodes | From treatment initiation (week 0) until end of treatment (up to 103 weeks)
  Measured as count of bleeds.
Arm 3: Number of treated traumatic bleeding episodes | From treatment initiation (week 0) until end of treatment (up to 103 weeks)
  Measured as count of bleeds.
Arm 3: Mim8 plasma concentration | From treatment initiation (week 0) until end of treatment (up to 103 weeks)
  Measured as µg/mL.
Arm 3: Device handling using haemophilia device assessment tool (HDAT) | At week 26 and week 52
  Measured as percentage of participants.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency dept. 2834, Study Director — Novo Nordisk A/S
Locations (137):
- United States (15):
  - Children's Hospital Los Angeles - Endocrinology, Los Angeles, California
  - UC Denver Hemoph & Thrombo Ctr, Aurora, Colorado
  - Univ of Miami/SCCC, Miami, Florida
  - St Joseph's Hospital Foundation, Tampa, Florida
  - Children's Healthcare Atlanta, Atlanta, Georgia
  - Rush University Med. Cntr, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Indiana Hemophilia-Thromb Ctr, Indianapolis, Indiana
  - University of Iowa_Iowa City, Iowa City, Iowa
  - Central Michigan University, Detroit, Michigan
  - Univ Hosp Cleveland Med Ctr, Cleveland, Ohio
  - Dayton Children Hemostati Ctr, Dayton, Ohio
  - Penn State MS Hershey Med Ctr, Hershey, Pennsylvania
  - St Christopher Hosp for Child, Philadelphia, Pennsylvania
  - Vanderbilt U Med Ctr_Nashville, Nashville, Tennessee
- Austria (2):
  - Universitätsklinik für Innere Medizin V, Innsbruck
  - AKH - Klin. Abt. f. Haematologie u. Haemostaseologie, Vienna
- Belgium (2):
  - Cliniques universitaires Saint-Luc - Service Hématologie, Brussels
  - UZ Leuven - Kindergeneeskunde, Leuven
- UMHAT Tsaritsa Yoanna - ISUL EAD, Pediatric clinical hematology and oncology, Sofia, Bulgaria
- Canada (2):
  - McMaster University, Hamilton, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
- China (13):
  - Beijing Children's Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Children's Hospital，Capital Medical University, Beijing, Beijing Municipality
  - Haemotology, Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - Nanfang Hospital, Southern Medical University-Haematology, Guangzhou, Guangdong
  - Tongji Hospital, Tongji Medical College of HUST-Hematology, Wuhan, Hubei
  - Tongji Hospital, Tongji Medical College of HUST, Wuhan, Hubei
  - Xiangya Hospital Central-South University, Changsha, Hunan
  - Jinan Central Hospital Affiliated to Shandong University, Jinan, Shandong
  - Jinan Central Hospital, Jinan, Shandong
  - Chengdu Women's and Children's Central Hospital, Chengdu, Sichuan
  - Institute of Hematology and Blood Diseases Hospital, Tianjin-Hematology, Tianjin, Tianjin Municipality
  - Children's Hospital, Zhejiang University School of Medicine-Hematology, Huzhou, Zhejiang
  - Jinan Central Hospital, Jinan
- Rigshospitalet - Department of Haematology, 2081, København Ø, Denmark
- France (4):
  - Hospices Civils de Lyon- Hopital Louis Pradel, Bron
  - Ap-Hp-Hopital de Bicetre-1, Le Kremlin-Bicêtre
  - Centre Hospitalier Universitaire de Lille-Institut Coeur Poumon, Lille
  - Centre Hospitalier Universitaire de Nantes-Hopital Hotel-Dieu, Nantes
- Germany (3):
  - Vivantes Netzwerk für Gesundheit GmbH - Vivantes Klinikum im Friedrichshain, Berlin
  - Universitätsklinikum Bonn - Institut für Experimentelle Hämatologie, Bonn
  - HZRM Haemophilie-Zentrum Rhein Main GmbH, Frankfurt am Main
- India (8):
  - Nirmal Hospital Pvt. Ltd., Surat, Gujarat
  - Seth GS medical college and KEM Hospital, Mumbai, Maharashtra
  - Sahyadri Clinical Research And Development Center, Pune, Maharashtra
  - Christian Medical College and Hospital, Ludhiana, Punjab
  - SMS Medical College & Hospital, Jaipur, Rajasthan
  - CMCV, Ranipet, Tamil Nadu
  - Post Graduate Institute of Child Health, Noida, Uttar Pradesh
  - Seth GS medical college and KEM Hospital, Mumbai
- St James's CRF, Dublin, Leinster, Ireland
- Sheba MC - The Israeli National Hemophilia Center, Tel Litwinsky, Israel
- Italy (9):
  - A.O.U. Policlinico Umberto I, Rome, Lazio
  - AOU Careggi Firenze, Florence
  - IRCCS Humanitas Research Hospital - Centro Trombosi e Malattie Emorragiche, Milan
  - Fondazione IRCSS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedaliera di Rilievo Nazionale Santobono Pausilipon, Napoli
  - Azienda Ospedaliera Santobono Pausilipon - U.S.D. Centro Regionale Pediatrico Malattie della Coagulazione, Napoli
  - Ospedale Pediatrico Bambino Ges, Roma
  - A.O.U. Policlinico Umberto I, Rome
  - A.O.U. Città della Salute e della Scienza di Torino-Ospedale, Torino
- Japan (9):
  - Nagoya University Hospital_Blood Transfusion, Aichi
  - Ota Memorial Hospital_Pediatrics, Gunma
  - Nara Medical University Hospital_Pediatrics, Nara
  - Saitama Children's Med Centre_Hematology-Oncology, Saitama
  - Jichi Medical University Hospital_Hematology, Tochigi
  - Jichi Medical University Hospital_Pediatrics, Tochigi
  - National Center for Child Health and Development_Hematology, Tokyo
  - Tokyo Medical Univ. Hospital_Laboratory Medicine, Tokyo
  - Ogikubo Hospital_Pediatries & Blood, Tokyo
- Latvia (2):
  - Stradini Clinic of Oncology, Riga
  - Children University Clinical Hospital, Riga
- Lithuania (2):
  - Vilnius University hospital Santaros klinikos, Vilnius
  - Centre of Oncology and Hematology, Vilnius University, Vilnius
- Malaysia (2):
  - Hospital Queen Elizabeth 1, Kota Kinabalu, Sabah
  - Hospital Ampang, Ampang, Selangor, Selangor
- Centro Multidisciplinario Para El Desarrollo Especializado De La Investigación Clínica En Yucatán S.C.P. (CEMDEICY S.C.P.), Mérida, Mexico
- Netherlands (2):
  - AmsterdamUMC AMC - Cardiologie, Amsterdam
  - UMC Utrecht, Van Creveldkliniek, Utrecht
- Poland (7):
  - Uniwersytecki Szpital Kliniczny W Poznaniu, Poznan, Greater Poland Voivodeship
  - Uniwersytecki Szpital Kliniczny im. J.Mikulicza-Radeckiego, Wroclaw, Lower Silesian Voivodeship
  - Instytut Hematologii i Transfuzjologii, Warsaw, Masovian Voivodeship
  - Intytut Hematologii i Transfuzjologii, Warsaw, Masovian Voivodeship
  - Szpital Uniwersytecki, Oddzial Kliniczny Hematologii, Krakow
  - Uniwersytecki Szpital Dzieciecy, Dzial Krwiolecznictwa, Lublin
  - Uniwersytecki Szpital Kliniczny im. J.Mikulicza-Radeckiego, Wroclaw
- Portugal (4):
  - Unidade Local de Saúde de Coimbra, E.P.E., Coimbra
  - Unidade Local de Saúde São José EPE- Hospital D. Estefânia, Lisbon
  - Centro Hospitalar Universitario De Santo Antonio E.P.E, Porto
  - Unidade Local de Saude de Sao Joao E.P.E, Porto
- Institut Oncologic "Prof. Dr. Ion Chiricuta" Cluj Napoca, Cluj-Napoca, Romania
- King Faisal Specialist Hospital & Research Centre, Riyadh, Riyadh, Saudi Arabia
- Serbia (2):
  - Clinical Centre of Serbia, Institute for Haematology, Belgrade
  - Clinical Centre of Vojvodina, Novi Sad
- Slovakia (3):
  - Univerzitna Nemocnica Martin, Martin
  - Vseobecna nemocnica Rimavska Sobota, Rimavská Sobota
  - Vranovska nemocnica, a.s., Vranov nad Topľou
- South Africa (2):
  - Wits Bara Clinical Trial Site, Johannesburg, Gauteng
  - Charlotte Maxeke Johannesburg Academic Hospital, Parktown, Johannesburg, Gauteng
- South Korea (4):
  - Daejeon Eulji Medical Center, Eulji University, Daejeon
  - Severance Hospital, Yonsei University Health System, Seoul
  - Gangdong Kyung Hee University Hospital, Seoul
  - Kyung Hee University Hospital at Gangdong, Seoul
- Spain (5):
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Sant Joan de Déu, Esplugues Llobregat
  - Hospital Universitario La Paz, Madrid
  - Hospital Carlos Haya, Málaga
  - Hospital Regional Universitario de Málaga, Málaga
- Switzerland (4):
  - Universitätsklinik für Hämatologie, Bern
  - Pädiatrische Onkologie-Hämatologie, Lucerne
  - Zentrum für Labormedizin, Sankt Gallen
  - Universitätsspital Zürich - Klinik für Medizinische Onkologie und Hämatologie, Zurich
- Taiwan (4):
  - Chung Shan Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital_main, Taipei
  - National Taiwan University Hospital, Taipei
- Turkey (Türkiye) (13):
  - Gazi University, Ankara, Beşevler/Ankara
  - Gazi Üniversitesi Hastanesi- Hematoloji, Ankara, Beşevler/Ankara
  - Istanbul University Oncology Institute, Capa-ISTANBUL, Capa-ISTANBUL
  - İstanbul Üniversitesi İstanbul Tıp Fakültesi Hastanesi- Onkoloji Enstitüsü, Capa-ISTANBUL, Capa-ISTANBUL
  - Akdeniz Üniversitesi Hastanesi- Hematoloji, Antalya, Konyaaltı/ Antalya
  - Acıbadem Adana Hastanesi-Hematoloji, Adana
  - Hacettepe Universitesi, Ankara
  - Hacettepe Üniversitesi Hastanesi- Hematoloji, Ankara
  - Akdeniz Universitesi, Antalya
  - Ege Universitesi Tip Fakultesi, Bornova-IZMIR
  - Ege Üniversitesi Hastanesi- Hematoloji, Bornova-IZMIR
  - Trakya University, Edirne
  - Trakya Üniversitesi Tıp Fakültesi Hastanesi-Hematoloji, Edirne
- United Kingdom (7):
  - Belfast City Hospital, Belfast
  - University Hospital of Wales - Haemophilia, Cardiff
  - Royal Free Haemophilia Comprehensive Care Center, London
  - Royal Free Hospital - Haemophilia, London
  - Evelina London Children's Hospital - Haemophilia, London
  - St Thomas' Hospital - Haemostasis and Thrombosis Centre, London
  - Royal Hallamshire Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com.
URL: http://novonordisk-trials.com